CLINICAL TRIAL: NCT00850486
Title: The Diagnostic Benefits of HyperQTM vs. Conventional ECG During Stress Test. A Comparison Study in Women Referred to Angiography.
Brief Title: Diagnostic Benefits of HyperQTM vs. Conventional ECG Stress Test. Comparison of HyperQ vs. Stress ECG in Women Before Angiography
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BSP Biological Signal Processing Ltd. (Industry)
Responsible Party: Professor Dan Tzivoni - Head of Cardiology Department, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: SHZ_02
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Ischemic Heart Disease
Keywords: women; ischemic heart disease; high frequency ECG; exercise stress testing; signal processing; ischemic heart disease in women
MeSH Terms: conditions — Myocardial Ischemia | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Exercise test with HyperQ technology — High frequency components of the QRS complex within the ECG signal are analyzed off-line to provide an indication of ischemia induced depolarization abnormalities

SUMMARY:
The purpose of this study is to verify the efficiency of the HyperQ technology compared with standard ECG analysis in detecting exercise induced ischemia in women who are referred to coronary angiography.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of mortality in women. In fact, CVD is responsible for a third of all deaths of women worldwide and half of all deaths of women over 50 years of age in developing countries. Historically, women have been underrepresented in clinical trials. The lack of good trial evidence concerning sex-specific outcomes has led to assumptions about CVD treatment in women, which in turn may have resulted in inadequate diagnoses and suboptimal management, greatly affecting outcomes. This knowledge gap may also explain why cardiovascular health in women is not improving as fast as that of men. Over the last decades, mortality rates in men have steadily declined, while those in women remained stable.

The treadmill exercise test is the classic initial investigation for the diagnosis of coronary artery disease (CAD), and significant ST depression on the ECG is the commonly used indicator of a positive test. Compared with men, in women it is known that ST depression is less likely to be associated with CAD. False positive rates of treadmill exercise testing have been reported to be as high as 67%, while positive predictive value is around 48-50%.

Coronary angiography is one of the most frequently performed procedures in women; however, non-obstructive (ie, <50% stenosis) CAD is frequently reported. Additionally, approximately 30% of women undergoing PTCA because of a positive exercise test are found to have normal coronary arteries. A successful outcome in the current study will significantly improve non-invasive diagnosis of CAD in women and may reduce the number of unnecessary invasive procedures performed.

ELIGIBILITY:
Inclusion Criteria:

* A woman who was referred to angiography.
* A woman who is able (i.e. no contraindications) to perform an exercise stress test
* A woman who signed an informed consent form.

Exclusion Criteria:

* Contraindications for an exercise test
* Wolff-Parkinson-White (pre-excitation) syndrome.
* Left Bundle branch block, Complete Right bundle branch block or QRS duration > 120 ms, change in QRS morphology during exercise
* Atrial Fibrillation or significant ventricular arrhythmia
* Treatment with Digoxin
* Pacemaker
* Having taken beta blockers within 24 hours before the exercise test
* Pregnancy or suspected pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-12 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
HyperQ results from the exercise test vs. angiography results | every 25 patients

CONTACTS AND LOCATIONS:
Overall Officials: Dan Tzivoni, Professor, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel